CLINICAL TRIAL: NCT06910111
Title: Cardio and Atherosclerosis Prevention and Treatment Via Fat Uptake REduction With a Specified Biopolymer: One Year Randomized Double-blind Placebo-controlled Clinical Investigation to Improve Vascular Health in Patients at Cardiovascular Risk: CAPTURE Study (Polyglucosamine for Cardio & Atherosclerosis Prevention and Treatment Via Fat Uptake REduction)
Brief Title: CAPTURE Study (Polyglucosamine for Cardio & Atherosclerosis Prevention and Treatment Via Fat Uptake REduction)
Acronym: CAPTURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Certmedica International GmbH (Industry)
Collaborators: Evidilya S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIV-IT-24-07-048534
Record Dates: First submitted 2025-02-27; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Atherosclerotic Disease
Keywords: CAPTURE formoline AtheroGuard

STUDY DESIGN:
Intervention Model Description: Two arms multicenter randomized double-blind placebo controlled clinical investigation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo consists of tablets
  Interventions: Device: Placebo
- Device (Experimental): 750 mg tablets main ingredient Polyglucosamin
  Interventions: Device: Polyglucosamine

INTERVENTIONS:
Device: Polyglucosamine — The treatment will continue for 12 months administering a customized Polyglucosamine (formoline AtheroGuard) (twice/day) before the two main meals for a total of 4 tabs/day (each tab consists of 750 mg). Controls will be conducted at screening/baseline, and after 3/6/9 and 12 months
  Arms: Device
Device: Placebo — 2x 2 Placebo tablets The treatment will continue for 12 months administering Placebo (twice/day) before the two main meals for a total of 4 tabs/day. Controls will be conducted at screening/baseline, and after 3/6/9 and 12 months
  Arms: Placebo

SUMMARY:
This clinical investigation is intended to confirm the application of a new intended purpose and a new indication for an already certified medical device. Therefore, it is a pivotal clinical investigation with a confirmatory type of design.

DETAILED DESCRIPTION:
Background and rationale The Investigational Product (formoline AtheroGuard, main ingredient: customized Polyglucosamine) administered by oral route before main meals binds fats in the stomach and intestine simply by physicochemical reaction and reduces their absorption and hydrolysis. The lower fat availability stimulates the mobilization of reserve lipids to be used for the metabolic processes and reduce the inflammatory cascade that can activate reactive cells (macrophages) in triggering atherosclerosis. Clinical data: Polyglucosamine treatment for 2 years significantly reduced Carotid Intima Media Thickness (CIMT). A recent meta-analysis has suggested a positive association between the progression of the Intima-Media Thickness (IMT) and cardiovascular risk. The results showed that interventional effects on the Carotid Intima-Media Thickness (CIMT) are also likely to reduce CV event rates.

Objective(s) The primary objective is to reduce or stabilize the increase of the arterial CIMT.

The reduction of plaque area, the change in plaques deposits, body weight, abdominal circumference, BMI, blood pressure, blood glucose, insulin resistance, insulin blood levels, hsCRP, oxidative stress, and the improvement of the lipid profile (reduction of triglycerides, total cholesterols, LDL and increase of HDL) are considered secondary objectives.

The safety objectives are to demonstrate the safety of formoline AtheroGuard 750 mg tablets administered for 12 months Design Two arms multicenter randomized double-blind placebo controlled clinical investigation

ELIGIBILITY:
Inclusion Criteria

* Outpatients of both genders, with CIMT > 1.00 mm suffering from hypertension and/or type II diabetes and/or hypercholesterolemia, under stable treatment for these conditions since at least 6 months.
* Age between 45-65
* BMI > 26 ≤35
* Total cholesterol ≥ 200 ≤ 240 mg/dL
* BP mm Hg: Mx ≥ 135 ≤ 160 ; Mn ≥ 75 ≤ 90 the subject must remain 10 min at rest in clinostatic position before measurement
* Blood glucose Mn ≥ 80 ; Mx ≤ 130 mg/dL
* The subjects suffering from hypertension, and/or diabetes, and/or hypercholesterolemia can be admitted provided that the diseases under chronic treatment are mitigated with no more than 2 drugs. By drug we mean any formulation (in tablets, capsules, fluid etc..) containing one or more active ingredients. This therapy has to be administered 4 hours before or after the product under evaluation.
* ESC score (European Society of Cardiology) < 10
* Informed consent must be obtained prior to participation.
* Subjects able to communicate adequately with the Investigator and to comply with the requirements for the entire study.
* Subjects must be willing and able to give informed consent/assent for participation in the study.
* Negative pregnancy test for women with childbearing capacity.

Exclusion criteria

* Age < 45 or > 65 years.
* Pregnancy or breastfeeding. During the study, women of reproductive age will have to use reliable contraceptive methods.
* Mx BP > 160 Mn > 90 despite a treatment of 6 months with common antihypertensive
* Total cholesterol > 240 mg/dL despite a treatment of 6 months with the common hypolipemic drugs
* Morning blood glucose > 130 mg/dL despite a treatment of 6 months with common oral hypoglycemic drugs
* BMI > 35
* ESC score (European Society of Cardiology) ≥ 10
* Myocardial infarction
* Neurological disorders
* Cancer
* Gout
* Kidney dysfunction (creatinine > 3 mg/dl)
* Liver dysfunction (ALT > 40 U/L)
* COPD (FEV < 80% of predicted value)
* Psychiatric diseases
* IBS
* Anemia (HB < 10 g/dl)
* Inability or unreliability of the Food Intake Assessment [4]
* Hypersensitivity to polyglucosamine
* Any medical condition or abnormality of clinical laboratory tests that needs systemic pharmacological treatment besides treatment for hypertension, type II diabetes or hypercholesterolemia. This means that local treatments will be allowed.
* Vulnerable subjects: incapacitated, immunocompromised, or other conditions which may bring to a condition of vulnerability.
* Subjects under emergency circumstances
* Treatment with orally applicable drugs exceeding application in the morning and in the late evening
* Current treatment with GLP-1 agonists, fosinopril, acarbose.
* In the case of treatment with food supplements the subject can be enrolled after 1 month of product withdrawal.
* Known allergy to crustaceans or one of the ingredients
* Chronic constipation
* Intestinal obstruction
* Intake of long-term medications that significantly slow down intestinal activity
* Current participation in any other investigational trials

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the reduction or stabilization of CIMT progression (measured through ultrasound) | Screening visit/baseline; after 6 months; after 12 months of treatment
  To demonstrate the benefit of formoline AtheroGuard reducing or stabilizing CIMT and plaques volume in patients suffering from dyslipidemia, hypertension, or type II diabetes.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Pisa University Hospital - Clinical Research Unit, Pisa, Tuscany
  - University Gabriele d'Annunzio Chieti - Pescara, Chieti
  - S. Maria della Misericordia Hospital, Perugia

IPD SHARING:
Plan to Share IPD: No